CLINICAL TRIAL: NCT06565208
Title: Phase 1, Randomized, Double-blind, Placebo-controlled, Staggered, Parallel, Single and Multiple Ascending Dose and Food Effect Study to Evaluate the Safety and PK of Oral SAT-3247 in Healthy Volunteers and Participants With DMD
Brief Title: First in Human SAD/MAD Safety and PK Study With Adult DMD Safety and PK Cohort
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Satellos Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SAT-3247-CL-101
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD; muscle regeneration
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Intervention Model Description: Single ascending dose cohorts and multiple ascending dose cohorts
Masking Description: Participants, Sponsor and Investigator are masked during Parts A-C. Part D is an open-label cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAT-3247 (Experimental): SAT-3247 is an oral tablet that is a potent, muscle penetrant, small molecule inhibitor of AAK1; inhibition of AAK1 rescues perturbed asymmetric division of satellite stem cells, resulting in increased muscle regeneration in animal models of DMD. In vitro and in vivo animal pharmacology studies have demonstrated the efficacy of SAT-3247 in improving muscle strength and the necessary target coverage to maximize functional muscle improvement.
  Part A: Participants will receive one oral dose of SAT-3247 in accord with cohort assignment (1) 10 mg, (2) 50 mg, (3) 150 mg, (4) 300 mg, (5) 400 mg Part B: Participants will receive one oral dose of SAT-3247 daily for seven days in accord with cohort assignment (1) 60 mg, (2) 120 mg, (3)180 mg, (4) 240 mg Part C: Participants will receive one oral dose of SAT-3247 150 mg, following completion of Part A at the same dose Part D: All participants will receive one SAT-3247 60 mg dose once daily for 5 consecutive days of each of 4 weeks
  Interventions: Drug: SAT-3247
- Placebo (Placebo Comparator): Part A: Participants will receive one oral dose of matched placebo in accord with cohort assignment of (1) 10 mg, (2) 50 mg, (3) 150 mg, (4) 300 mg, (5) 400 mg Part B: Participants will receive one oral dose of matched placebo daily for seven days in accord with cohort assignment (1) 60 mg, (2) 120 mg, (3)180 mg, (4) 240 mg Part C: Participants will receive one oral dose of matched placebo 150 mg, following completion of Part A at the same dose
  Interventions: Drug: matched placebo

INTERVENTIONS:
Drug: SAT-3247 — SAT-3247 is an oral tablet that is a potent, muscle penetrant, small molecule inhibitor of AAK1; inhibition of AAK1 rescues perturbed asymmetric division of satellite stem cells, resulting in increased muscle regeneration in animal models of DMD. In vitro and in vivo animal pharmacology studies have demonstrated the efficacy of SAT-3247 in improving muscle strength and the necessary target coverage to maximize functional muscle improvement.
  Other Names: SAT3247; AAK1 inhibitor
  Arms: SAT-3247
Drug: matched placebo — matched placebo
  Other Names: placebo
  Arms: Placebo

SUMMARY:
This is a first-in-human (FIH), Phase 1 study of orally administered SAT-3247 in healthy adult volunteers (HVs) and adult participants with DMD to determine safety, tolerability, pharmacokinetics and pharmacodynamics.

DETAILED DESCRIPTION:
This is a first-in-human (FIH), Phase 1 study of orally administered SAT-3247 in healthy volunteers (HVs) and adult participants with DMD. The study will be conducted in 4 parts.

Part A is a Single Ascending Dose (SAD) part that will enroll approximately 40 HVs in up to 5 dose cohorts. Each participant will receive a single oral dose of SAT 3247 or matched placebo on Day 1; each cohort will receive a higher dose than the prior cohort. Part B is a Multiple Ascending Dose (MAD) part that will enroll approximately 32 HVs in up to 4 sequential dose cohorts. Each participant will receive a daily oral dose of SAT-3247 or matched placebo on Day 1 to Day 7 each cohort will receive a higher dose than the prior cohort. Part C will assess the effect of food on the PK of SAT-3247 in a fixed sequence, crossover design. The dose to be tested will be determined by the Safety Review Committee (SRC) following review of safety, tolerability, and available PK and PD data from Part A. Approximately 8 healthy participants who completed Part A at the anticipated dose level (in a fasted state) will crossover into a subsequent fed cohort and receive a single dose of the same randomized IP at the same dose level that they received in Part A but, following a high fat meal. Part D is a open-label Multiple Dose cohort that will comprise 10 adult males with genetically confirmed DMD. Each participant will receive SAT-3247 once daily for 5 consecutive days of each of 4 weeks

ELIGIBILITY:
Parts A-C enroll healthy volunteers; only entry criteria for Part D are described below.

Part D Inclusion Criteria:

* Able and willing to provide written informed consent after the nature of the study has been explained and prior to the commencement of any study procedures.
* Considered reliable and capable of adhering to the protocol and able and willing to attend the necessary visits to the study site according to the judgment of the PI or designee.
* Male patients ≥18 to ≤ 40 years (inclusive at the time of informed consent), or considered an adult able to consent to participate in a clinical study in the jurisdiction in which the study is being conducted.
* Non-smoker and must not have used any tobacco or cannabis products within 2 months prior to Screening.
* Has a definitive diagnosis of DMD based on documented clinical findings and prior genetic testing with a confirmed mutation in the DMD gene.
* BMI ≥ 18.0 kg/m2 and ≤ 32.0 kg/m2 and weight ≥ 50 kg at Screening.
* Stable dose of systemic glucocorticosteroids, heart medications, and/or other supportive medications, vitamins and supplements according to the standard of care for DMD for 3 months prior to the Screening visit and for the duration of the study. Participants that are not receiving glucocorticosteroids are also eligible, but must refrain from initiating glucocorticosteroid treatment for the duration of the trial.
* Agree to abstain from donating blood or blood products during the study and for up to 3 months after the administration of the IP.

Part D Exclusion Criteria:

* Underlying psychological condition or history of any mental illness that, in the opinion of the PI or designee, would make it unlikely for the participant to comply with the protocol or complete the study per protocol.
* Presence of acute or chronic illness or history of chronic illness sufficient to invalidate the patient's participation in the study or make it unnecessarily hazardous in the judgment of the PI.
* Any clinically significant medical, surgical, or psychiatric abnormality that, in the judgment of the Investigator, is likely to interfere with study compliance, the safe participation of the subject or the assessment of safety or efficacy.
* Any surgical procedures (eg, stomach bypass) or medical condition that might affect absorption of medicines.
* Has donated blood within 60 days of IP administration or donated plasma within 7 days of IP administration or experienced loss of blood ≥500 mL within 2 months of IP administration.
* Fever (body temperature >38°C) or symptomatic viral or bacterial infection within 2 weeks prior to Screening.
* Poor pill swallowing ability as determined by PI.
* Presence or history of severe allergic or anaphylactic reactions, or sensitivity to the IP or its constituents.
* History of relevant atopy including any confirmed significant allergic reactions against any drug, or multiple drug allergies (non-active hay fever is acceptable).
* History of malignancy, except for non-melanoma skin cancer excised more than 2 years prior to Screening and cervical intraepithelial neoplasia that has been successfully cured more than 5 years prior to Screening.
* Abnormal ECG findings at Screening and or Day -1 that are considered by the PI or designee to be clinically significant.
* QT value, measured at Screening visit, greater than 450 msecs (male) on 12-lead ECG, using Fridericia's formula (QTcF) for correction.
* Pulse ≤ 45 or ≥ 100 beats per minute (bpm); systolic blood pressure ≤ 90 mmHg or ≥ 160 mmHg, or diastolic blood pressure ≤ 50 mmHg or > 95 mmHg at Screening.
* History or presence of a condition associated with significant immunosuppression.
* History of life-threatening infection (eg, meningitis).
* Infections requiring parenteral antibiotics within 6 months prior to Screening.
* Positive test for hepatitis C antibody (HCV), hepatitis B surface antigen (HBsAg), human immunodeficiency virus (HIV) antibody.
* Vaccination with a vaccine within 28 days prior to the first administration of IP.
* Creatine kinase > ULN or ALP, AST, bilirubin, and/or ALT >1.5 × ULN at Screening.
* Anticipated change to prescription medication, over the counter medications, vitamins, supplements, and/or herbal remedies during the course of the trial.
* Anything that the PI or designee considers would jeopardize the safety of the participant, prevent complete participation in the study (including the possibility that the participant will not cooperate with the requirements of the protocol) or compromise interpretation of the study data.
* An employee, consultant, and/or immediate family member (ie, first degree relative, spouse, adoptees, or legal dependents) of the site, Sponsor, or the CRO.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — adult DMD patients assigned male at birth
Enrollment: 77 (Actual)
Dates: Start 2024-08-21 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent adverse events | Part A: Day 1-3; Part B: Day 1-8; Part C: Day 1-3; Part D: Day 1-28
  Safety and tolerability of SAT-3247 as compared to placebo

SECONDARY OUTCOMES:
Serum plasma Pharmacokinetics of SAT-3247 | Part A: Day 1-3; Part B: Day 1-8; Part C: Day 1-3; Part D: Day 1-28
  Plasma PK parameters including Cmax, Tmax, AUC, terminal half-life, CL/F, Vz/F, and ratios of Cmax and AUC

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - CMAX, Adelaide, South Australia
  - Veritus, Bayswater, Victoria

IPD SHARING:
Plan to Share IPD: No